CLINICAL TRIAL: NCT01879124
Title: Correlation Between Renal Vascular Resistive Index, Renal Allograft Histology and Outcome
Brief Title: Resistive Index Measurements After Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Maarten Naesens, Prof. Dr. Maarten Naesens, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: KidneyTX-UZLEUVEN-RI
Record Dates: First submitted 2013-06-10; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kidney transplant recipients: All de novo renal allograft recipients transplanted at the University Hospitals Leuven between March 2004 and October 2007

SUMMARY:
The purpose of this study is to evaluate the prognostic performance of intrarenal resistive index in the first years after kidney transplantation on graft function and on patient and graft survival. In addition, the determinants of the intrarenal resistive index, including a detailed analysis of the relation between graft histology and the intrarenal resistive index, will be assessed.

DETAILED DESCRIPTION:
Since March 2004, and as part of routine clinical practice, protocol renal allograft biopsies are routinely performed at implantation and at 3, 12 and 24 months after transplantation, in all patients who receive a kidney transplant at the University Hospitals Leuven, unless there is a medical contra-indication or patient refusal to undergo this procedure. The biopsies are scheduled using a dedicated Microsoft Access database ("Biopsy Database"), that is maintained on the central servers of the University Hospitals Leuven. Patients who have an unexplained change in renal allograft function, undergo additional clinically indicated indication biopsies. These biopsies are also recorded in the aforementioned Microsoft Access Database.

All clinical data, including pretransplant donor and recipient characteristics, and post-transplant follow-up data are directly stored and maintained in a prospectively collected electronic database (CCL database until 06/2012, transferred to the central KWS database in 2012). This electronic database is the only existing clinical database for these patients, and contains all clinical patient charts. No written records are collected.

All renal allograft biopsies will be rescored by a single renal pathologist according to the most recent Banff classification, blinded for the clinical parameters and timing of the biopsy. These rescoring data are directly entered in the dedicated Microsoft Access database ("Biopsy Database").

Just prior to performing a renal allograft biopsy with ultrasound guidance, and as part of the routine clinical procedure, duplex measurements are performed by the radiologist who will perform the biopsy. The peak systolic velocity (Vmax) and the minimal diastolic velocity (Vmin) are determined in each patient in two to three representative interlobar arteries. The resistive index is calculated as [1 - (V min/V max)]. This procedure is repeated at three different places in the kidney (lower, interpolar and upper pole). These data are directly entered in the central electronic clinical database system (KWS, see above).

All electronic data will be transferred to a SAS database at time of data extraction.

ELIGIBILITY:
Inclusion Criteria:

Single kidney transplantation

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All de novo renal allograft recipients transplanted at the University Hospitals Leuven between March 2004 and October 2007
Sampling Method: Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2004-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Overall renal allograft survival | 7 years after transplantation
Death-censored graft survival | 7 years after transplantation
Patient survival | 7 years after transplantation
Reduction of 50% or more in the eGFR from the value measured at the time of ultrasonography | 7 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Naesens, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Naesens M, Heylen L, Lerut E, Claes K, De Wever L, Claus F, Oyen R, Kuypers D, Evenepoel P, Bammens B, Sprangers B, Meijers B, Pirenne J, Monbaliu D, de Jonge H, Metalidis C, De Vusser K, Vanrenterghem Y. Intrarenal resistive index after renal transplantation. N Engl J Med. 2013 Nov 7;369(19):1797-806. doi: 10.1056/NEJMoa1301064. PMID 24195547